CLINICAL TRIAL: NCT07271992
Title: TREND-02 - a Phase II Exploratory De-escalation Trial of Neoadjuvant Sacituzumab Govitecan Plus Tislelizumab (SG/I) in Early Triple-negative Breast Cancer
Acronym: TREND-02
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Collaborators: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Yingying Xu, Professor, First Hospital of China Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y-2024-PT-0285
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: TNBC, Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SG+I (Experimental): SG 10mg/kg， d1,d8 q3w
  + I 200mg, d1 q3w 6 cycles （18 weeks）
  Interventions: Drug: SG+I

INTERVENTIONS:
Drug: SG+I — SG 10mg/kg， d1,d8 q3w + I 200mg, d1 q3w 6 cycles （18 weeks）

SUMMARY:
Refining neoadjuvant chemoimmunotherapy and establishing predictive biomarkers remain pivotal challenges in early TNBC. Although SG/I (sacituzumab govitecan/PD-1 inhibitor) shows clinical promise, validation of responder identification tools is warranted. This phase II trial aims to identify a precision TNBC population suitable for de-escalated neoadjuvant therapy with sacituzumab govitecan plus tislelizumab, based on differential Trop-2 expression (±) and PD-L1 status (CPS >10% vs. <10%). Primary endpoints include pCR rate and safety; exploratory biomarker analyses will assess mechanisms of response/resistance

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years; 2. Histologically confirmed stage II or III primary invasive TNBC TNBC defined as: immunohistochemistry (IHC) ER and PR <1%; HER2-negative, IHC 0 or 1+, IHC 2+, ISH-; 3. ECOG performance status score 0-1; 4. Provision of an acceptable tumor sample prior to randomization; 5. Bone marrow hematopoietic and organ function must meet study requirements; Without growth factor support or blood transfusion, ANC ≥ 1.5 × 10⁹/L, platelets ≥ 100 × 10⁹/L, hemoglobin ≥ 9 g/dL; Bilirubin ≤ 1.5 × upper limit of normal (ULN); ALT and AST ≤ 2.5 × ULN; Creatinine ≤ 1.5 × ULN; Urinalysis showing proteinuria < 2+ or 24-hour urine protein < 1 g; Coagulation function must be normal, defined as: International Normalized Ratio (INR) and/or Prothrombin Time (PT) ≤ 1.5 × ULN and/or Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN. If anticoagulant therapy is ongoing, PT must remain within the therapeutic range for the anticoagulant used.

Serum amylase ≤ 1.5×ULN and serum lipase ≤ 1.5×ULN.

Exclusion Criteria:

* 1. Evidence of severe/uncontrolled systemic disease, including active infections requiring intravenous therapy, severe chronic gastrointestinal disease associated with diarrhea, active bleeding disorders, severe cardiac or psychiatric disorders, or history of allogeneic organ transplantation; 2. History of other primary malignancies with known active disease within 3 years prior to randomization and low potential for recurrence (excluding adequately excised non-melanoma skin cancers and treated carcinoma in situ); 3. Active or documented history of autoimmune or inflammatory diseases; 4. Presence of distant metastases; 5. Active or uncontrolled hepatitis B or C infection, uncontrolled HIV infection, or active tuberculosis; 6. History of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy, any clinically active interstitial lung disease, or immune-related pneumonitis induced by immunotherapy; 7. Any prior or concurrent surgery, radiotherapy, or systemic anticancer therapy for TNBC; 8. Prior exposure to the following treatments: Immunosuppressive drug therapy within 14 days before the first study intervention Live attenuated vaccines within 30 days before the first study intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2030-12-14 (Estimated); Study Completion 2031-12-14 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) rate | From enrollment to the end of treatment at 24 weeks
  To evaluate the pathological complete response (pCR) rate (ypT0/Tis ypN0) following neoadjuvant sacituzumab govitecan plus immunotherapy (SG/I) in biomarker-selected TNBC